CLINICAL TRIAL: NCT02902380
Title: The Effect of Dexmedetomidine on Neuroendocrine Stress Hormone Release and Heart Rate Variability in Patients Undergoing Major Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 4-2016-0644
Record Dates: First submitted 2016-09-06; First posted 2016-09-15 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine Group (Experimental): dexmedetomidine infusion (0.4 mcg/kg/h) from immediately after anesthetic induction to end of surgery
  Interventions: Drug: dexmedetomidine group
- Control Group (Placebo Comparator): 0.9% saline infusion
  Interventions: Drug: control group

INTERVENTIONS:
Drug: dexmedetomidine group — dexmedetomidine infusion (0.4 mcg/kg/h) from immediately after anesthetic induction to end of surgery
  Arms: Dexmedetomidine Group
Drug: control group — 0.9% saline infusion
  Arms: Control Group

SUMMARY:
Surgical stress induces stress hormone release and sympathetic hyperactivation. Dexmedetomidine has sympatholytic effect and attenuates stress responses. This study investigate the effect of dexmedetomidine on stress responses and autonomic nervous system balance in patients undergoing major spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* patient between 20 and 70 of age with ASA physical status Ⅰ-Ⅲ
* patient scheduled for major spine surgery

Exclusion Criteria:

* ASA physical status Ⅳ
* congestive heart failure
* severe hepatorenal disease
* insulin dependent DM(diabetes mellitus)
* cancer or metastasis
* pregnancy
* problem with communication

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Stress hormone level | immediately after anesthetic induction
  The levels of stress hormone including epinephrine, norepinephrine, cortisol, and glucose will be measured during spinal surgery.
Stress hormone level | 1 hour after start of surgery
  The levels of stress hormone including epinephrine, norepinephrine, cortisol, and glucose will be measured during spinal surgery.
Stress hormone level | 2-hour after start of surgery
  The levels of stress hormone including epinephrine, norepinephrine, cortisol, and glucose will be measured during spinal surgery.
Stress hormone level | 1 second after the end of surgery
  The levels of stress hormone including epinephrine, norepinephrine, cortisol, and glucose will be measured during spinal surgery.
Stress hormone level | 1 hour after the end of surgery
  The levels of stress hormone including epinephrine, norepinephrine, cortisol, and glucose will be measured during spinal surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No